CLINICAL TRIAL: NCT01577524
Title: The Use of Diluted Povidone Iodine Irrigation in Spine Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: We had very low recruitment rates that would have resulted in several years being added to the study to achieve an appropriate sample size.
Sponsor: Attabib, Najmedden, M.D. (Individual)
Responsible Party: Principal Investigator, Dr. Najmedden Attabib, Principle Investigator, Attabib, Najmedden, M.D.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2009-1350
Record Dates: First submitted 2012-03-30; First posted 2012-04-16 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Povidone-Iodine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diluted Povidone Iodine Solution (Active Comparator)
  Interventions: Drug: Povidone-Iodine
- Normal Saline Wash (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Povidone-Iodine — Subjects in the treatment group will receive 3.5% diluted Povidone Iodine solution in the surgical incision in a quantity sufficient to fill the wound to the level of the skin. The Povidone Iodine solution will be maintained in the incision for 3 minutes, after which it will be flushed from the wound with normal saline solution.
  Other Names: Betadine
  Arms: Diluted Povidone Iodine Solution
Drug: Saline — Subjects in the Placebo Comparator group will receive normal saline solution in a quantity sufficient to fill the wound to the level of the skin. The saline solution will be maintained in the incision for 3 minutes, after which it will be flushed from the wound with additional saline solution to replicate the saline wash procedure followed in the Treatment group.
  Arms: Normal Saline Wash

SUMMARY:
The purpose of the study is to determine whether diluted Povidone Iodine solution used to irrigate surgical wounds during spine surgery decreases the incidence of surgical site infections.

DETAILED DESCRIPTION:
Post-operative infections in spine surgery have been extensively investigated in the literature. These investigations focus on the efficacy of using peri-operative antibiotics, Povidone Iodine skin preparations, the effects of shaving around the surgical sit, and the use of intra-operative diluted Povidone Iodine wound irrigation in preventing post-operative infections.

Povidone-iodine is a complex of polyvinyl pyrrolidine and tri-iodine ions widely used as an antiseptic agent. It has bactericidal activity against a wide spectrum of pathogens, including methicillin-resistant Staphylococcus aureus (MRSA). The safety of its use intra-operatively has been evaluated in animal studies and also supported through Randomized Controlled Trials in spinal surgery and in other surgical subspecialties.

The purpose of this study is to evaluate the efficacy of the intra-operative use of diluted Povidone Iodine solution in reducing post-operative infections when used for irrigating surgical incisions during spinal surgery compared with 0.9% Sodium Chloride Irrigation Solution (i.e. normal saline solution).

The primary outcome measure will be seen as a reduction in the number of post-operative infections. As a result and although not directly measured, it is suspected that a reduction in post-operative infections may result in quicker healing with fewer complications and pain.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-75
* Undergoing posterior surgical spinal procedure for degenerative spine disease, extra-dural tumors, trauma, or spinal deformity
* No obvious potential infective focus
* Patient willing to enroll

Exclusion Criteria:

* Age <18 or >75
* Identified infective focus in the body, including furuncles,or acne at surgical incision site
* Patient with discitis or spinal osteomyelitis
* Dural tear
* Potential use of Bone Morphogenic Protein (BMP)
* Iodine hypersensitivity
* Out of province patients due to difficulty in arranging follow up visits
* Minimal invasive spine surgical procedure (MISS) due to difficulty of having diluted Betadine solution contact soft tissue with the use if MISS retractors
* Pregnancy
* Inability to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of post-operative infections diagnosed in both treatment and control groups | Twelve months post operation
  The Centers for Disease Control (CDC)definition of surgical site infections (SSI)will be used for this study.This definition addresses both superficial and deep surgical site infections.
  Outcome will be determined by the number of superficial, deep, and total (superficial plus deep) wound infections for each group.

CONTACTS AND LOCATIONS:
Overall Officials: Najmedden Attabib, MD, Principal Investigator — Neurosurgery Department, Saint John Regional Hospital
Locations (1):
- Saint John Regional Hospital, Saint John, New Brunswick, Canada

REFERENCES:
- [Background] Celik SE, Kara A. Does shaving the incision site increase the infection rate after spinal surgery? Spine (Phila Pa 1976). 2007 Jul 1;32(15):1575-7. doi: 10.1097/BRS.0b013e318074c39f. PMID 17621202
- [Background] Cheng MT, Chang MC, Wang ST, Yu WK, Liu CL, Chen TH. Efficacy of dilute betadine solution irrigation in the prevention of postoperative infection of spinal surgery. Spine (Phila Pa 1976). 2005 Aug 1;30(15):1689-93. doi: 10.1097/01.brs.0000171907.60775.85. PMID 16094267
- [Background] Georgiade G, Riefkohl R, Georgiade N, Georgiade R, Wildman MF. Efficacy of povidone-iodine in pre-operative skin preparation. J Hosp Infect. 1985 Mar;6 Suppl A:67-71. doi: 10.1016/s0195-6701(85)80048-7. PMID 2860178
- [Background] Goldenheim PD. In vitro efficacy of povidone-iodine solution and cream against methicillin-resistant Staphylococcus aureus. Postgrad Med J. 1993;69 Suppl 3:S62-5. PMID 8290460
- [Background] Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG. CDC definitions of nosocomial surgical site infections, 1992: a modification of CDC definitions of surgical wound infections. Infect Control Hosp Epidemiol. 1992 Oct;13(10):606-8. No abstract available. PMID 1334988
- [Background] Rubinstein E, Findler G, Amit P, Shaked I. Perioperative prophylactic cephazolin in spinal surgery. A double-blind placebo-controlled trial. J Bone Joint Surg Br. 1994 Jan;76(1):99-102. PMID 8300691
- [Background] Schubert R. Disinfectant properties of new povidone-iodine preparations. J Hosp Infect. 1985 Mar;6 Suppl A:33-6. doi: 10.1016/s0195-6701(85)80043-8. PMID 2860173
- [Background] Sindelar WF, Brower ST, Merkel AB, Takesue EI. Randomised trial of intraperitoneal irrigation with low molecular weight povidone-iodine solution to reduce intra-abdominal infectious complications. J Hosp Infect. 1985 Mar;6 Suppl A:103-14. doi: 10.1016/s0195-6701(85)80054-2. PMID 2860153
- [Background] Strohecker J, Piotrowski WP, Lametschwandtner A. The intra-operative application of povidone-iodine in neurosurgery. J Hosp Infect. 1985 Mar;6 Suppl A:123-5. doi: 10.1016/s0195-6701(85)80057-8. PMID 2860156
- [Background] Wilson AP, Treasure T, Sturridge MF, Gruneberg RN. A scoring method (ASEPSIS) for postoperative wound infections for use in clinical trials of antibiotic prophylaxis. Lancet. 1986 Feb 8;1(8476):311-3. doi: 10.1016/s0140-6736(86)90838-x. PMID 2868173
- [Background] Fang A, Hu SS, Endres N, Bradford DS. Risk factors for infection after spinal surgery. Spine (Phila Pa 1976). 2005 Jun 15;30(12):1460-5. doi: 10.1097/01.brs.0000166532.58227.4f. PMID 15959380
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716